CLINICAL TRIAL: NCT03573661
Title: A Pilot Multi-Institutional Study to Evaluate the Accuracy of a Breast Cancer Locator in Patients With Palpable Cancers
Acronym: BCL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Richard J. Barth,Jr., MD, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: D16196
Record Dates: First submitted 2018-06-19; First posted 2018-06-29 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Palpable Breast Cancer
Keywords: Breast Conserving Surgery; Breast Imaging; Breast Cancer Locator; Supine MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Breast Cancer Locator (BCL) (Experimental): The Breast Cancer Locator (BCL) uses 3D printing to create a bra-like plastic form that matches the breast surface when the patient is in the supine MRI (and surgical) position. This locator will be constructed pre-operatively, sterilized and provided to the surgeon at the time of procedure.
  Interventions: Device: Breast Cancer Locator (BCL)

INTERVENTIONS:
Device: Breast Cancer Locator (BCL) — This locator will be constructed pre-operatively, sterilized and provided to the surgeon at the time of procedure. The outline of the breast cancer on the breast surface at the point where the cancer is closest to the skin is built into the locator, so that the surgeon can simply apply the locator to the patient's breast and trace the tumor outline on the skin.

SUMMARY:
The project objective is to determine whether the Breast Cancer Locator (BCL) can safely and effectively localize breast cancers in patients treated at locations distant from the site of BCL manufacture. This information will be transmitted to CairnSurgical, Inc. where the BCL will be fabricated, tested for quality assurance, sterilized and shipped to the patient's surgeon. The surgeon will then utilize the BCL at the time of resection of the palpable breast cancer.

DETAILED DESCRIPTION:
The primary purpose of the study is to determine whether a device called the Breast Cancer Locator (BCL) accurately identifies the location of cancer in the breast. The Breast Cancer Locator is a plastic bra-like form that gives the surgeon information about the location of the cancer in the breast. The location information is derived from an MRI which is obtained with the patient lying flat on their back (just as they are on an operating room table). The BCL is then custom-made for the patient using 3D printing technology.

The surgeon can feel the cancer, and the surgeon will remove the cancer by feeling the edges of it as the surgeon would normally. Since the cancer can be felt, the surgeon does not need an image guidance system such as the BCL to locate the cancer in the breast. Other women may have breast cancers that cannot be felt, but are only identified by mammography or MRI. If the BCL proves to accurately localize breast cancer, it may be a useful guide for the surgeon for these other women.

Additionally, the investigators want to determine whether this technology can be successfully employed at multiple sites and what, if any, complications occur during surgery as a result of using this device. The BCL has been used in 19 patients at Dartmouth with no complications.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Histologic diagnosis of palpable invasive breast cancer or ductal carcinoma in situ.
3. Patient desire to undergo breast surgery (lumpectomy or non-skin sparing mastectomy).
4. Ability to voluntarily provide informed consent to participate prior to any study-related assessments/procedures being conducted.
5. The cancer enhances on prone breast MRI imaging
6. The cancer is visible on mammography.

Exclusion Criteria:

1. Absolute contraindication to MRI, including presence of implanted electrical device (pacemaker or neurostimulator), aneurysm clip, or metallic foreign body in or near eyes.
2. Severe claustrophobia.
3. Contraindication to use of gadolinium-based intravenous contrast, including life- threatening allergy or compromised renal function (creatinine > 2.0).
4. History of median sternotomy.
5. Pregnancy. Patient attestation that they are not pregnant will be acceptable.
6. Patients receiving neoadjuvant chemotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who had the localization wire placed within the cancer on the specimen mammogram | Within approximately 60 Days post-surgery (all measures are collected by the time of patient follow-up visit within approximately 60 days after surgery, and recorded by the surgeon and radiologist in Case Report Forms (CRF forms).
  Yes/No answer from Radiologist. Final measure will be % of cases rated Yes (wire deployed within the cancer on specimen mammogram).

SECONDARY OUTCOMES:
Whether the study Radiologist can accurately define boundaries of the tumor from the supine MRI images | Within approximately 60 days following surgery
  Yes/No answer from Radiologist. Final measure will be % of cases rated Yes (tumor segregated accurately from supine MRI). The data is recorded by the radiologist on the CRF form.
Time from supine MRI to delivery of the Breast Cancer Locator (BCL) device to the surgeon | Within approximately 60 days following surgery
  Unit of measure is in days. Final measure will be average days to delivery among all patients. The data is recorded by the surgeon on the CRF form.
Whether the BCL allowed the surgeon to successfully mark in/on the breast skin surface the items he or she needs to see during the surgery, including tumor edges and locations where wires will be placed | Within approximately 60 days following surgery
  Yes/No answer from Surgeon. Final measure will be % of cases rated Yes (BCL enabled surgeon to successfully place all cues). The data is recorded by the surgeon on the CRF form.
Lumpectomy specimen volumes | Within approximately 60 days following surgery
  Unit of measure is in mL, calculated by water displacement. Final measure will be average volume (mL) among all patients. The data is recorded by the study sponsor, Cairn Surgical, on the CRF form.
Operative times (Average time per operation) | Within approximately 60 days following surgery
  Unit of measure is in minutes. Final measure will be average operative time (min.) among all patients. Data is collected by the surgeon from operative notes and placed in the CRF form.
The tumor margins, which the pathologist measures (as the distance from the tumor to the specimen edge) | Within approximately 60 days following surgery
  Unit of measure is in cm. Final measure will be average margin (in cm) among all patients. Data is collected by the surgeon from the pathology report and reported in the CRF form.
Complications from surgery | Within approximately 60 days following surgery
  Surgeon to list any complications - which could include infections or bruising. Final measure will be % of patients with complications. Data is collected from the surgeon either post-operatively, if there were operative complications; or at the post-operative follow-up appointment with the patient, if she reports any complications then. It is also possible this data could be collected at any time between surgery and follow up appointment by the patient calling the surgeon's office to report it. The surgeon records this data in the CRF form.
Surgeon satisfaction with the technical aspects of surgery guided by the Breast Cancer Locator | Within approximately 60 days following surgery
  Yes/No answer. Final measure will be % of surgeons who say Yes to satisfaction with the procedure. Data is collected from the surgeon and reported in the CRF form.

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Barth, Jr., MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (4):
- United States (4):
  - Lahey Hospital & Medical Center (Lahey Clinic), Burlington, Massachusetts
  - Cheshire Medical Center, Keene, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - St. Joseph Hospital, Nashua, New Hampshire